CLINICAL TRIAL: NCT07387094
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Study to Assess the Efficacy and Safety of XW003 Injections in Obese Participants With Obstructive Sleep Apnea But Not Receive Positive Airway Pressure Therapy
Brief Title: A Study of XW003 in Obese Participants With Obstructive Sleep Apnea But Not Receive Positive Airway Pressure Therapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCW0502-5031
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: OSA - Obstructive Sleep Apnea; Obesity
Keywords: XW003; Ecnoglutide; Obesity; OSA; GLP-1
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XW003 Injection (Experimental): once weekly
  Interventions: Drug: XW003 injection
- Placebo (Placebo Comparator): once weekly
  Interventions: Drug: placebo with matching volume

INTERVENTIONS:
Drug: XW003 injection — subcutaneous injection
  Arms: XW003 Injection
Drug: placebo with matching volume — subcutaneous injection
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the efficacy and safety of XW003 injections in obese participants with OSA but not receiving PAP

DETAILED DESCRIPTION:
In this Phase III study, eligible participants will be randomized into one of the two cohorts in a 1:1 ratio to receive once-weekly subcutaneous XW003 injection or placebo, including a dose-escalation period, for up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 28.0 kg/m2;
2. The results of PSG meet the diagnosis criteria of OSA and with an AHI ≥15 at screening;
3. Participants must not have used PAP for at least 4 weeks prior to screening and not use PAP during the study;
4. Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

1. History of endocrine disorders which have significant impact on body weight;
2. Diagnosis of diabetes (except gestational diabetes), ketoacidosis or hypertonic state/coma;
3. HbA1c ≥6.5% at screening;
4. Fasting blood glucose ≥7.0 mmol/L or 2-hour blood glucose ≥11.1 mmol/L after oral glucose tolerance test (OGTT) at screening; participants with FBG ≥6.1 mmol/L but <7.0 mmol/L require OGTT;
5. Have diagnosis of Cheyne Stokes Respiration, or diagnosis of Central or Mixed Sleep Apnea with % of mixed or central apneas/hypopneas ≥50%;
6. Respiratory and neuromuscular diseases that could interfere with the results of the trial;
7. Diagnosis of Obesity Hypoventilation Syndrome or daytime hypercapnia;
8. Change of body weight >5% within 3 months prior to screening (self-reported);
9. Have a prior or planned surgical treatment for obesity (except liposuction or abdominoplasty if performed more than 1 year prior to screening);
10. Have received any medication for body weight loss and blood glucose lowering or medication that could lead to significant body weight increase, within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2027-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Apnea-Hypopnea Index (AHI) | at week 48

SECONDARY OUTCOMES:
Percent Change From Baseline in AHI | at week 48
Percentage of Participants With ≥50% AHI Reduction From Baseline | at week 48
Percentage of Participants With AHI <5 or With AHI 5-14 With Epworth Sleepiness Scale (ESS) ≤10 | at week 48
Percent Change From Baseline in Body Weight | at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Dr, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No